CLINICAL TRIAL: NCT01148342
Title: Neurobiology and Pharmacokinetics of Acute MDMA Administration
Brief Title: Neurobiology and Pharmacokinets of Acute MDMA Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: 999904394; 04-DA-N394
Record Dates: First submitted 2010-06-19; First posted 2010-06-22 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-07-18

CONDITIONS: Substance-Related Disorders
Keywords: Ecstacy; fMRI; Alternative Matrices; Cognitive Training; Brain Imaging
MeSH Terms: conditions — Substance-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine

INTERVENTIONS:
Drug: MDMA
Drug: (+/-)3,4-methylenedioxymethamphetamine Hydrochloride, MDMA HCI Capsules — 0, 1.0 & 1.6 mg/kg

SUMMARY:
Background:

* 3,4-Methylenedioxymethamphetamine (MDMA), commonly known as ecstasy, is a synthetic psychoactive drug that has shown a steep increase in recreational use and abuse by young people in recent years. Research studies have reported that chronic MDMA users who also consume other legal and illegal substance show memory deficits; however, because of the combination of drugs often involved, it is difficult to determine MDMA s contribution to these effects.
* Only a few studies have examined the immediate physical and behavioral effects of MDMA given at dose levels commonly used in young adults. Researchers are interested in using functional magnetic resonance imaging (fMRI) to examine changes in brain activity and function in MDMA users compared with users of other drugs and non-drug-using individuals.

Objectives:

- To evaluate the effects of MDMA on thinking and brain function.

Eligibility:

- Individuals between 18 and 30 years of age who are (1) current users of MDMA (2), current drug users who do not use MDMA, or (3) healthy non-drug-using volunteers.

Design:

* Participants will complete one training session and three scanning sessions.
* Before the start of the study, participants will complete questionnaires about medical and psychological history, and provide information about past or current drug use. Researchers will introduce the tasks to be performed during the scanning session(s), and will allow participants to practice the tests.
* Participants will provide urine, saliva, and hair samples for testing before the start of the study, and multiple times during each scanning session.
* Participants who use MDMA and participants who use other drugs will stay overnight at the clinical center prior to each scanning session. Participants who do not use drugs can spend the night prior to scanning or arrive at the clinical center on the morning of the scanning session.
* Participants who use MDMA will receive either MDMA or a placebo during the scanning sessions, and will not be told which one they have received. Because of the nature of MDMA, participants will be required to stay at the clinical center until the effects of the drug have worn off, and will be required to return to the clinical center on the following day for a follow-up examination.
* During the study, participants will be asked to do one or more tasks selected by the researchers. The tasks will be performed on a computer in an MRI machine, and may involve receiving monetary rewards for actions, memory and reaction-time tests, or other tests that involve responding to instructions on the screen.

DETAILED DESCRIPTION:
Background: 3,4-Methylenedioxymethamphetamine (MDMA), commonly known as ecstasy, is a synthetic compound that has shown a steep increase in abuse by young people in recent years. In animals, when high and multiple doses of MDMA were given, serotonergic toxicity was observed. Clinically, the number of severe ecstasy related acute toxicities is low in relation to the extent of recreational use. Data from some retrospective studies report memory deficits in abstinent chronic users who often abuse MDMA with other illicit and licit substances; therefore, it is difficult to determine MDMA s contribution to observed cognitive deficits. There are few prospective controlled MDMA human administration studies that describe its acute physiological and behavioral effects following doses commonly used in young adults. We propose a functional magnetic resonance imaging (fMRI) study to examine specific changes in brain activity and cognitive performance and to correlate these changes with plasma MDMA concentrations.

Goals: The primary goals are identification of MDMA effects on human brain function and elucidation of the relationship of effects to plasma MDMA concentrations. We propose a within-subject design of changes in memory, attention, affect, semantic processing and decision-making performance following placebo and two recreational MDMA doses with simultaneous fMRI monitoring and plasma collections. Secondly, pharmacokinetic data will be collected on the disposition of MDMA and metabolites in plasma, urine, oral fluid, sweat, breath, and hair. These data are needed to accurately interpret drug concentrations in alternative biological matrices in order for drug tests to function as a deterrent to drug use in drug abuse treatment, law enforcement, military, and workplace drug testing programs. Pharmacokinetic data will also enable drug tests to serve as valid diagnostic tools in emergency medicine and public safety settings, as well as useful objective outcome measures in treatment research.

Subject Population: Eighteen current MDMA users will complete the neurocognitive and pharmacokinetics group. Thirty-six MDMA non-using controls will include 18 non-drug using participants and 18 drug using (primarily cannabis) participants. Controls in each group will be matched to MDMA users in the neurocognitive and pharmacokinetics group. All participants must be between the ages of 18 and 40. The estimated target enrollment, based on ecstasy use by race/ethnic group and Baltimore demographics, will be 41% female and 59% male, 83% Caucasian, 14% African American, 3% Asian, and 2% Hispanic.

Experimental Design and Methods: A randomized, balanced, double blind, within-subject drug administration study with placebo, low (1.0 mg/kg, approximately 70 mg) and high (1.6 mg/kg, approximately 112 mg) doses of MDMA is proposed. The non-drug using and drug using control groups will be matched to MDMA users in the neurocognitive and pharmacokinetics group for sex, age, IQ, education level and intersession interval. The drug using control group will control for cannabis and other drug usage in the MDMA group. The drug using control group is necessary because many MDMA users also use other drugs, primarily cannabis. Control groups allow for a between-subjects analysis for trait differences between the population groups, as well as provide normative data for the cognitive tasks. Drug using control group participants will stay on the clinical research unit overnight prior to each of the three sessions; non-drug using control group participants will arrive the morning of each session. Participants from the MDMA group will complete three separate stays, each lasting approximately 26 hours, within one year. While under the influence of MDMA, qualified participants will perform memory, attention, semantic processing, affect and decision-making tasks before, during, and after fMRI scanning. Physiological, behavioral and biochemical measures of all MDMA users will be monitored throughout the study to determine onset, magnitude and duration of pharmacodynamic effects. Blood, urine, oral fluid, sweat, breath, and hair specimens will be collected from MDMA users for analysis of MDMA and metabolite concentrations by GC/MS and/or LC/MS/MS to determine the disposition and pharmacokinetics of MDMA.

Risks and Benefits: A main potential risk of this study is associated with acute cardiovascular responses to MDMA administration; however, these doses have proven safe and well tolerated in previous human studies conducted within the US and abroad. In addition, impaired cognitive function has been reported following long-term MDMA use in some but not all studies. A potential benefit of the proposed study is to understand how MDMA affects human brain function at doses employed by recreational users. Additionally, advances will be made in understanding MDMA pharmacokinetics.

ELIGIBILITY:
* INCLUSION CRITERIA: Participants must:

  1. Be between the ages of 18 and 40.
  2. If MDMA group, have consumed at least five tablets of ecstasy in their lifetime with no clinically significant adverse medical or psychiatric reactions from using the drug or other stimulants and must have used at least once within the past 30 days (Drug Use Survey), with no current intention to stop MDMA use. History of ecstasy consumption is supported by a minimum of one positive urine amphetamines or hair MDMA drug test within the past 90 days. Urine drug tests at scanning visits must not be positive for drugs, other than amphetamines and cannabis. Scanning visits can be rescheduled once due to a positive urine test for other drugs.
  3. If control group, have no history of MDMA use (Drug Use Survey) and have negative urine test for amphetamines. If in the non-drug using group, must have a negative urine test for non-therapeutic psychoactive drugs at screening and scanning visits. Lifetime cannabis use for these participants cannot exceed ten times, with no use in the past two years (Timeline Follow-Back Method (146)). At screening, drug using controls may test positive for other drugs, other than amphetamines. At scanning, drug using controls may be positive for cannabis only. Scanning visits can be rescheduled once due to a positive urine test for other drugs.
  4. Be without current clinically significant medical problems that would preclude safe study participation.
  5. If female, must use a reliable method of birth control or abstain from sexual intercourse. Female participants will be counseled that a urine pregnancy test cannot detect pregnancies within 7 to 14 days of conception.
  6. Have an 8th grade reading and comprehension level.

     Additional requirements for participants undergoing neurocognitive testing:
  7. Have an IQ ? 85 determined by the Wechsler Abbreviated Scale of Intelligence (WASI) (The Psychological Corporation, 1999).
  8. Be right handed (Edinburgh Handedness Inventory (147)).
  9. Speak English as their first language.

EXCLUSION CRITERIA: Participants must NOT:

1. Have known major medical or axis I psychiatric diagnosis other than substance abuse (Structured Clinical Interview (SCID) for the Diagnostic & Statistical Manual of Mental Disorders IV (DSM-IV) criteria). Participants with a history of psychotropic medicine use will be evaluated by the MRP on a case-by-case basis to uncover the precise diagnosis for the use of the drug. Individuals who have substance dependence other than nicotine or cannabis, based on DSM IV criteria, will be excluded from the study. Prospective participants will be excluded if they smoke more than two packs of cigarettes per day.
2. If MDMA user, be currently using (within 30 days of MDMA administration) one of the following inhibitors of CYP2D6 or CYP3A4 or inducers of CYP3A4:

   CYP2D6 inhibiting drugs<TAB><TAB><TAB><TAB>

   Antidepressants: paroxetine, fluoxetine, sertraline, fluvoxamine, nefazodone, venlafaxine, clomipramine, amitriptyline, citalopram, bupropion

   Antipsychotics: haloperidol, perphenazine, thioridazine, levomepromazine, pimozide, fluphenazine

   Antiarrythmics: quinidine

   Protease inhibitors: ritonavir

   CYP3A4 inhibiting drugs

   Antidepressants: nefazodone, fluvoxamine, fluoxetine, sertraline, paroxetine, venlafaxine, norfluoxetine

   Azole antifungals: ketoconazole, itraconazole, fluconazole

   Protease inhibitors: ritonavir, nelfinavir, amprenavir

   Nonnucleoside reverse transcriptase inhibitors: efavirenz, delavirdine

   Histamine H2 -receptor antagonists: cimetidine

   Macrolide antibiotics: clarithromycin, erythromycin

   Calcium channel blockers: diltiazem

   In addition, participants will be advised to limit their consumption of grapefruit juice.

   CYP3A4 inducing drugs

   Antibacterials: rifampin

   Antidepressants: St. John s wart

   Anticonvulsants: carbamazepine, phenobarbital, phenytoin

   Adrenocortical steroids: dexamethasone

   If potential participants need to continue taking these drugs as part of a physician prescribed treatment regimen, they will be excluded for safety purposes. Potential participants will be advised that there should be a minimum 30-day abstention from the use of these listed compounds prior to MDMA administration.
3. If MDMA user, SBP greater than 135 and DBP greater than 85 taken after at least 5 minutes rest, tachycardic (resting HR greater than 100 bpm), or hypercholesterolemic (total cholesterol greater than 250 mg/dL) if above the age of 30.
4. If MDMA user, have hemoglobin levels less than 12.5-g/100 mL if male and less than 12-g/100 mL if female.
5. If MDMA user, have clinically significant abnormal resting 12-lead ECG.
6. If female, be pregnant or nursing.
7. Have liver function tests greater than 3 times upper limit of normal range.
8. Be unable to comply with task demands.
9. Have a history of neurological illnesses including but not limited to stroke, central nervous system tumor, encephalitis or other CNS infection, multiple sclerosis or other demyelinating diseases, epilepsy, movement disorders, or migraine headaches severe enough to require treatment.
10. If non-drug using control, have a hair test positive for non-therapeutic psychoactive drugs.
11. If drug using control, have hair test results that are inconsistent with self-reported drug use.

    Additional exclusion criteria for participants undergoing neurocognitive testing:
12. <TAB>Have head trauma with loss of consciousness for greater than 3 minutes
13. <TAB>Have a positive HIV serology test (retested after six months).
14. <TAB>Have an ADHD Screening Rating Scale score greater than or equal to 24 on either the A or B subscale.
15. <TAB>Have a positive Fluorescent Treponemal Antibody Absorption Test (FTA-ABS) confirmatory test for syphilis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2004-02-10; Study Completion 2012-07-18 (Actual)

PRIMARY OUTCOMES:
MDMA effects on human brain function and relationship between plasma MDMA concentrations and human brain function.

SECONDARY OUTCOMES:
MDMA pharmacokinetics in various biological matrices.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huestis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Pentney AR. An exploration of the history and controversies surrounding MDMA and MDA. J Psychoactive Drugs. 2001 Jul-Sep;33(3):213-21. doi: 10.1080/02791072.2001.10400568. PMID 11718314
- [Background] Rosenbaum M. Ecstasy: America's new "reefer madness". J Psychoactive Drugs. 2002 Apr-Jun;34(2):137-42. doi: 10.1080/02791072.2002.10399947. PMID 12691203
- [Background] Greer GR, Tolbert R. A method of conducting therapeutic sessions with MDMA. J Psychoactive Drugs. 1998 Oct-Dec;30(4):371-9. doi: 10.1080/02791072.1998.10399713. PMID 9924843